CLINICAL TRIAL: NCT01551485
Title: Postoperative Sleep Disturbances After Zolpidem Treatment in Fast-track Hip and Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lene Krenk, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: H-3-2011-022
Record Dates: First submitted 2012-02-06; First posted 2012-03-12 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Sleep Duration on the First Night After Surgery
MeSH Terms: interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zolpidem (Experimental)
  Interventions: Drug: Zolpidem
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zolpidem — The effect of Zolpidem 10 mg for the first night after surgery is asssessed using PSG
  Arms: Zolpidem
Drug: Placebo — Pacebo tablet, blinded given on the first night after surgery
  Arms: Placebo

SUMMARY:
Sleep after surgery has been found to be very distrubed immediately after major surgery. This is also seen after fast-track hip and knee replacement with length of stay of less than 3 days. Disturbed sleep has many adverse effects i.e. fatigue, possible hyperalgesia and decline in cognitive abilities.

ELIGIBILITY:
Inclusion Criteria:

* Total hip or knee replacement in fast-track setup
* Age 60 years or above
* ASA class 1-3

Exclusion Criteria:

* Anesthesia within the pas 30 days
* Daily use of alcohol > 21 units / week
* Use of anxiolytics or hypnotics within the past 30 days
* Inability to read and understand Danish
* Marked reduction of sight or hearing
* Parkinson's disease or other neurological disaese causing function deficits
* Inability to cooperate to sleep monitoring
* allergy to the drug tested

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Change in sleep time on the first postoperative night compared to preoperatively. | first night postoperatively - 24 hours
  The primary endpoint is an evaluation of sleep stages on the first night postoperatively compared to preoperative measures for the same individual

CONTACTS AND LOCATIONS:
Overall Officials: Lene Krenk, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Gentofte Hospital, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Krenk L, Jennum P, Kehlet H. Postoperative sleep disturbances after zolpidem treatment in fast-track hip and knee replacement. J Clin Sleep Med. 2014 Mar 15;10(3):321-6. doi: 10.5664/jcsm.3540. PMID 24634631